CLINICAL TRIAL: NCT01851460
Title: Radiofrequency Ablation (RFA) for the Treatment of Liver Abscesses in Patients With Chronic Granulomatous Disease
Brief Title: Radiofrequency Ablation for Liver Abscesses From Chronic Granulomatous Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI choose to close the study
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130117; 13-I-0117
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2019-10

CONDITIONS: Chronic Granulomatous Diseases (CGD) and Liver Lesions
Keywords: Non-surgical Liver Lesions; Chronic Granulomatous Disease (CGD); Microorganisms; Bacteria; Liver Lesions
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA (Experimental): All subjects enrolled onto this study will receive treatment of their liver abscess (es) by RFA ablation
  Interventions: Device: Cool-tip RF Ablation System

INTERVENTIONS:
Device: Cool-tip RF Ablation System — RFA therapy will be administered according to the instructions of the RFA device manufacturer. After infiltration of the skin (for percutaneous approach) with a local anesthetic, the needle probe will be directed into the lesion. For all methods, the needle placement is confirmed to be within the lesion by ultrasound or other imaging modality as appropriate. After confirming needle placement, the lesion will be heated to a target temperature of >75 (Infinite)c for up to 15 minutes. The exposure time may be varied depending on the temperatures achieved. Depending on the size of the lesion to be ablated, multiple passes of the probe as well as multiple ablation cycles may be performed. Adequacy of ablation will be monitored by ultrasound throughout the procedure. Depending on the size of the lesions and the time required to complete the ablation, multiple lesions may be treated as staged procedures so as to improve safety.

SUMMARY:
Background:

- Abscesses are a pocket of infection in an organ or tissue. Patients with a disease called chronic granulomatous disease (CGD) often develop these abscesses. CGD is an inherited disorder that affects how white blood cells function. Liver abscesses in people with CGD often require surgery to remove them and treat the infection. However, some people with CGD cannot have full surgery because it would be too risky. Researchers want to try a procedure called radiofrequency ablation (RFA) to treat these liver abscesses. RFA can usually be done without a major operation. This study will see if RFA is a safe and effective treatment for liver abscesses in patients with CGD.

Objectives:

- To see if RFA is a safe and effective treatment for CGD-related liver abscesses.

Eligibility:

- Individuals between 18 and 75 years of age with CGD who have liver abscesses that cannot be treated with surgery.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies will be performed on the liver.
* Participants will have RFA for the abscesses. RFA is an image-guided technique that heats and destroys specific tissue, such as tumor tissue. It will target any abscesses on the liver.
* After the procedure, participants will stay in the hospital for monitoring before being released.
* Participants will have regular follow-up visits for up to 1 year after treatment. Blood and urine samples will be collected. Additional imaging studies will be performed.

DETAILED DESCRIPTION:
Radiofrequency Ablation (RFA) has become an increasingly common therapeutic treatment for neoplasms in the liver. A number of devices are now Food and Drug Administration cleared for this indication, and a growing body of literature supports this technique as a therapeutic option for patients with primary or metastatic hepatic malignancies. In vivo animal studies have also shown that this technique can also be used to treat infections. Insertion of the thermal energy delivery probe into an infected liver abscess destroys the bacteria while preserving surrounding tissue. Off-label use of RFA was successfully used to treat 22 abscesses in 4 patients with chronic granulomatous disease who had inoperable liver abscesses. The proposed clinical trial will specifically evaluate the feasibility, safety, and to a lesser extent, efficacy of RFA to treat liver abscesses in subjects with previously diagnosed chronic granulomatous disease. This will be a non-randomized case study conducted at the Clinical Center at the National Institutes of Health. One RFA device will be used. Ten subjects will be enrolled. If the method proves to be both feasible and safe, detailed analysis on efficacy will be performed. RFA eventually could play an important clinical role in patients with chronic granulomatous disease and liver abscesses that are not amenable to surgical management and are without other effective therapeutic options, or might otherwise be incompletely treated with surgical resection and debridement alone.

ELIGIBILITY:
* INCLUSION/ELIGIBILITY CRITERIA:

A patient will be included if he or she meets all of the following criteria:

1. Has documented chronic granulomatous disease
2. Age 18 - 75
3. Has a liver abscess infected with Staphylococcus aureus or other microorganism susceptible to RFA, but is not an optimal candidate for curative surgical resection either due to location of disease, multiplicity of disease, or previous surgery or other comorbidities, such as pulmonary insufficiency, or has other contraindications to general anesthesia or perioperative management or refuses surgery.
4. Is willing to return to NIH for imaging scans
5. Is willing to undergo testing or procedures associated with this protocol
6. Has failed long term antibiotic treatment and abscess drainage if applicable.

EXCLUSION CRITERIA:

A patient will be excluded if he or she satisfies 1 or more of the following criteria:

1. Positive results for toxin-producing bacteria obtained from liver biopsy in the pertinent abscess.
2. Is a good candidate for liver-curative open surgical resection and does not refuse the surgery.
3. Is not a candidate for RFA therapy due to lesion size or location.
4. Has a prothrombin time (PT) or partial thromboplastin time (PTT) >1.5 times normal (except in patients who have a known lupus anticoagulant or other condition which a hematologist deems will not cause excessive bleeding despite the abnormal coagulation parameters).
5. Has a platelet count <50,000/mm(3) which cannot be maintained despite platelet transfusions.
6. If you are pregnant.
7. Any condition that, in the investigator s opinion, places the patient at undue risk by participating in the study

Please Note: Co-morbidities in critically ill patients will not themselves constitute exclusion criteria because the cause of their illness/condition may require the use of RFA as a less invasive treatment than surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Safety of RFA in the treatment of liver abscesses in CGD subjects | Fater each patient completes the study
  The primary objective of this study is to determine the safety of radiofrequency ablation (RFA) in the treatment of liver abscesses in subjects with chronic granulomatous disease (CGD).

SECONDARY OUTCOMES:
Determine if RFA is a reasonable treatment options | After last patient completes the study
  To determine if RFA is a reasonable treatment option for patients with liver abscesses who are not suitable candidates for completely curative hepatic surgery
Compare recovery outcomes | After last patient completes the study
  To compare the recovery outcomes of patients undergoing RFA versus historical controls for patients undergoing surgery for treatment of liver abscesses

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Livraghi T. Radiofrequency ablation, PEIT, and TACE for hepatocellular carcinoma. J Hepatobiliary Pancreat Surg. 2003;10(1):67-76. doi: 10.1007/s10534-002-0714-y. PMID 12918460
- [Background] Lublin M, Bartlett DL, Danforth DN, Kauffman H, Gallin JI, Malech HL, Shawker T, Choyke P, Kleiner DE, Schwartzentruber DJ, Chang R, DeCarlo ES, Holland SM. Hepatic abscess in patients with chronic granulomatous disease. Ann Surg. 2002 Mar;235(3):383-91. doi: 10.1097/00000658-200203000-00010. PMID 11882760
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-I-0117.html